CLINICAL TRIAL: NCT06136845
Title: The Correlation Between Microbiome of Esophageal Cancer Patients and Post Esophagectomy Anastomotic Leaks
Acronym: microbiome
Status: Recruiting | Type: Observational
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, Irit Ben-Aharon MD, Oncology Division head, Rambam Health Care Campus
Other Study IDs: 0672-19-RMB
Record Dates: First submitted 2023-11-06; First posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Esophageal Tumors
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- non anastomotic leak: Non anastomotic clinical leak'
- anastomotic clinical leak: anastomotic clinical leak'

SUMMARY:
Esophageal cancer continues to be one of the most challenging topics and the subjects of numerous studies. Surgery is the mainstay for curative treatment and the need to improve all aspects of perioperative management in order to reduce morbidity and mortality, continues to be of immense importance.

Cited as the sixth most common cause of cancer-related death worldwide, esophageal cancer has a distinct geographic distribution known as the esophageal cancer belt: north central China through the central Asian republics to northern Iran, and from eastern to southern Africa.

Squamous-cell carcinoma and adenocarcinoma are the two main histological subtypes of esophageal cancer, in a geographic differentiation as well, with squamous-cell carcinoma as the most common esophageal cancer subtype worldwide. Though adenocarcinoma is at a considerable rise in Western populations and has become the predominant subtype North America, Australia and Europe.

Although an ongoing improvement has been marked in the long-term survival after esophagectomy, it is still a highly invasive procedure with serious post-operative complications and entails a high morbidity and mortality rates.

Rates of mortality and morbidity range vastly in the literature with 30-day mortality reaching 11-22%. Complication rates up to 50%, with anastomotic leaks as the main complication ranging widely 0-35%.

Various risk factors have been proposed as contributors to mortality and morbidity in general and to anastomotic leaks in particular. These include both patient and tumoral characteristics such as premedical history and perioperative factors as tumor location, surgical technique and perioperative treatment.

The microbiome as a contributor to a patients' disease progression and management is of great interest in the understanding and better management of cancer patients as a whole and of the gastrointestinal tract in specific.

The contribution of the microbiome of a patient to colorectal cancer progression and to anastomotic leaks in the post-operative period has been addressed vastly in the literature in recent years, showing a distinct correlation to specific microbiota profile. Shogan et al. depicted a potential molecular mechanism of bacterial-driven anastomotic leak. It was shown that strains of the commensal organism Enterococcus faecalis could cause anastomotic leakage by causing direct collagen degradation at the site of a freshly constructed anastomosis, and indirectly by bacterial-induced over activation of host matrix metalloproteinase 9 (MMP9).

A geographic differentiation in microbiota of Colorectal Cancer (CRC) was also shown by comparing tumor tissue and adjacent tissue of Colorectal Cancer patients from the US and Spain, elaborating yet another aspect of the importance of microbiome of cancer patients.

Oropharyngeal microbiome profiling has been proven as a possible predictor for post esophagectomy pneumonia projecting on overall survival as well.

A recent study by Rishindra et al from the university of Michigan shows a strong correlation of post esophagectomy anastomotic leaks and increased bacterial variance in preoperative oral and gastric flora.

We hypothesize that a correlation exists between microbiome of esophageal cancer patients and post esophagectomy anastomotic leaks.

According to former evidence microbiota are integrated into the tumor and therefore the microbial profile of the host (patient) may be represented by tumor microbiota.

In this proposed study, we intend to characterize retrospectively the microbial signature of esophageal tumors and to study whether there is a correlation between differential microbial signature and risk of post esophagectomy anastomotic leaks.

ELIGIBILITY:
Inclusion Criteria:

* Cancer patients who have a surgery sample at Rambam Pathology Department
* Given written informed consent to Rambam BioBank or Midgam for collection, storage, collection of information and use for future research
* Patients with non-metastatic esophageal cancer (mid/Siewert 1/Siewert 2) who developed esophageal leak
* Patients with non-metastatic esophageal cancer (mid/Siewert 1/Siewert 2) who had no post-op complication.

Exclusion Criteria:

• Patients who had complete response are excluded due to lack of tumoral tissue in the specimen for analysis

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with esophageal tumors
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-01-13 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
To evaluate a correlation between microbial signature of esophageal cancer and post esophagectomy anastomotic leaks | All through the trial, On average 36 months.
  To evaluate a correlation between microbial signature of esophageal cancer and post esophagectomy anastomotic leaks
To assess the possibility of mapping a specific microbiota profile as a risk factor for anastomotic leaks | All through the trial, On average 36 months.
  To assess the possibility of mapping a specific microbiota profile as a risk factor for anastomotic leaks
To characterize the microbiota of esophageal cancer patients differentiating it by: - demographic criteria - tumor characteristics | All through the trial, On average 36 months.
  To characterize the microbiota of esophageal cancer patients differentiating it by:
  * demographic criteria
  * tumor characteristics

CONTACTS AND LOCATIONS:
Overall Officials: Irit Ben Aharon, MD, Principal Investigator — Rambam Health Care Campus
Locations (1):
- Rambam Health Care Campus, Haifa, Israel